CLINICAL TRIAL: NCT03565276
Title: Tranexamic Acid for Prevention of Postpartum Haemorrhage: a Dose-finding Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Sinai Health System (Other); University of Toronto (Other); University of Waterloo (Other); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Rohan D'Souza, Maternal-Fetal Medicine Physician, Mount Sinai Hospital, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-0001-A (MSH-REB)
Record Dates: First submitted 2018-04-23; First posted 2018-06-21 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Post Partum Hemorrhage
Keywords: Post partum hemorrhage; Tranexamic acid; TXA; Dose-finding; Prevention
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: As part of the dose-escalation design, the investigators will start with 5mg/kg, half the smallest described dose, on a sample of up to 5 women. They will continue to administer TxA doses in increments of 5mg/kg to each successive batch of 5 women. If the number of treatment successes cannot statistically rule out a value < 75% (< 4 of 5 women are successes due to values in the low range), the dose will be increased by 5mg/kg for the next set of 5 women, and so on, until a maximum dose of 30mg/kg is reached, a dose deemed safe based on earlier studies in different populations. Once treatment success is determined at a certain dose, i.e. 4/5 women have levels in the therapeutic range), a total of 20 women will be administered that dose to ensure that 75% i.e. 18/20 women are successes at that dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: TXA (Experimental): Intravenous Tranexamic Acid beginning at 5mg/kg administered as part of a dose-escalation design.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — A single dose of intravenous TxA in 100ml of 0.9% sodium chloride at 50mg/min, via a dose-escalation design
  Other Names: TxA; Cyklokapron

SUMMARY:
Published trials on tranexamic acid (TxA) for prevention have used a variety of fixed (0.5gm or 1gm) and body-weight adjusted (10mg/kg or 15mg/kg) doses of TxA. Given the wide range of bodyweights of pregnant women in contemporary obstetric practice, it is critical to determine the minimum effective dose of TxA, so as to avoid under- or over-dosing. The rationale of this study is to determine the minimum effective dose of TxA that is required to attain therapeutic plasma levels of TxA, established at 5-15mg/L, following administration of a single dose of intravenous (IV) TxA after childbirth and the clamping the umbilical cord, and before delivery of the placenta. Following birth of the infant, and upon clamping the umbilical cord, the investigators will administer a single dose of IV TxA in 100ml of 0.9% sodium chloride at 50mg/min according to the dose-escalation schedule described below. The slow rate of infusion has been chosen to prevent untoward effects such as hypotension that have been noted when the rate of infusion has exceeded 100mg/min. As part of the dose-escalation design, the investigators will start with 5mg/kg, half the smallest described dose, on a sample of up to 5 women. They will continue to administer TxA doses in increments of 5mg/kg to each successive batch of 5 women. If the number of treatment successes cannot statistically rule out a value < 75% (< 4 of 5 women are successes due to values in the low range), the dose will be increased by 5mg/kg for the next set of 5 women, and so on, until a maximum dose of 30mg/kg is reached, a dose deemed safe based on earlier studies in different populations. Once treatment success is determined at a certain dose, i.e. 4/5 women have levels in the therapeutic range), a total of 20 women will be administered that dose to ensure that 75% i.e. 18/20 women are successes at that dose.

DETAILED DESCRIPTION:
Research question: What is the minimum effective dose required for attainment of therapeutic plasma levels of 5-15mg/L in postpartum women?

Study design: Pharmacokinetic study using a dose-escalation design.

Trial treatment and dosage regimen: Following recruitment and prior to the caesarean delivery, the anaesthesiologist will insert a large-bore cannula into the participant's antecubital vein and draw blood for a complete blood count (CBC), which will be used in tandem with 24-hour post-delivery CBC to estimate blood loss, and serum creatinine to rule out elevated serum creatinine levels, a study exclusion criterion. Following birth of the infant, and upon clamping the umbilical cord, the anaesthesiologist will administer a single dose of IV TxA in 100ml of 0.9% sodium chloride at 50mg/min according to the dose-escalation schedule described below. All participants will receive oxytocin 20 international units (IU) IV in 1 litre of 0.9% sodium chloride at the rate of 125 ml/hour with placental delivery, as part of active management of the third stage of labour.

Endpoints Primary endpoints - Plasma levels of TxA: These will be obtained via serial blood draws at baseline (before TxA administration), and at 15, 30, 60 minutes and 120 minutes after administration of TxA, (as its maximum effect is within the 60 minutes and therapeutic plasma concentrations are maintained for 7-8 hours after administration). Blood will be drawn at baseline (before administration of TxA) in order to confirm zero plasma levels of TxA, as part of quality assurance. Blood will be collected in a standard citrate tube (Vacutainer, NJ, USA), centrifuged soon after collection and the plasma (supernatant) stored at -80°C before analysis. TxA will be extracted from plasma using solid phase microextraction, and concentrations measured using tandem liquid chromatography/mass spectrometry.

Secondary endpoints: (a) Total blood loss in 24 hours following childbirth will be determined by the reference standard methods - direct measurement (blood collected in suction apparatus) and gravimetric (weighing of linen) and by using formulae to determine blood loss using pre- and post-delivery haemoglobin and haematocrit as we have previously described (b) Early adverse events will be recorded prior to discharge and delayed events will be obtained at the six-week postpartum visit or via phone call.

Expected duration of subject participation, duration of all trial periods and follow up: The intervention will only be administered once, and blood drawn at baseline and 15, 30, 60 and 120 minutes after administration, as described above. Again, as described above, data on early adverse events will be collected prior to discharge from hospital and those on delayed adverse events will be obtained at the time of the routine 6-week postpartum visit in person or via a telephone interview. There will be no additional follow up.

Stopping rules: As the drug will be administered as a slow infusion in the operating room, it will be stopped immediately if any adverse events are noted. Thereafter, no further drug will be administered, and therefore stopping rules do not apply. Participants will be allowed to withdraw from the study at any point without affecting their clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or greater
* Pregnant with a single fetus
* Undergoing planned caesarean delivery for a non-medical indication
* ≥ 37 completed weeks of gestation

Exclusion Criteria:

* Contraindications to use of TxA (i.e. acute arterial/venous thrombosis, hypersensitivity to TxA, history of seizures, moderate to severe renal failure from any condition, defective colour vision, subarachnoid haemorrhage and disseminated intravascular coagulation (abnormally increased activation of pro-coagulant pathways))
* Medical conditions that could influence bleeding and/or the pharmacokinetics of TxA (i.e. personal/family history of bleeding disorders, receipt of warfarin seven days or heparin 24 hours prior to caesarean delivery, hypertensive disorders of pregnancy, need for intra- or post-operative blood transfusions and postpartum thromboprophylaxis)
* Women with morbidly adherent placentae scheduled for planned caesarean-hysterectomies
* Use of concomitant medications that could result in drug interactions (hydrochlorothiazide, desmopressin, sulbactam-ampicillin, carbazochrome, ranitidine or nitroglycerin)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Plasma levels of TxA | 0, 15, 30, 60, 120 minutes
  Measured in mg/L. The 3 samples drawn at 15, 30 and 60 minutes should be between 5-15mg/L to be considered treatment success. Levels at 0 minutes is expected to be zero and 120 minutes expected to be sub-therapeutic.

SECONDARY OUTCOMES:
Early Adverse events | maximum 24 hours
  Having experienced any one of the following: nausea/vomiting, abdominal pain, diarrhoea, disturbed color vision, skin rash, headache, migraine, nasal/sinus symptoms, musculoskeletal/back pain, joint pains, muscle cramps, fatigue, anorexia, dizziness, seizures, blood clots or low blood pressure between delivery and discharge from hospital.
Early adverse event 2 - Ga | six weeks
  Having experienced any one of the early adverse outcomes described above between discharge from hospital and the six-week postpartum visit

CONTACTS AND LOCATIONS:
Overall Officials: Rohan D'Souza, Principal Investigator — Rohan.Dsouza@sinaihealthsystem.ca
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No